CLINICAL TRIAL: NCT05987943
Title: Lecturer of Oral and Maxillofacial Surgery
Brief Title: A Pedicled Buccal Periosteal Flap for the Closure of Oro-antral Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marwa Taha Ibrahim (Other)
Responsible Party: Sponsor-Investigator, Marwa Taha Ibrahim, principle investigator, Tanta University
Organization: Tanta University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-OS-9-22-6
Record Dates: First submitted 2023-07-14; First posted 2023-08-14 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Oroantral Fistula
Keywords: oroantral fistula; A Pedicled Buccal Periosteal Flap
MeSH Terms: conditions — Oroantral Fistula

STUDY DESIGN:
Intervention Model Description: patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healing.recurrence of oroanral fistula (Other): A Pedicled Buccal Periosteal Flap for the Closure of Oro-antral Fistula
  Interventions: Procedure: A Pedicled Buccal Periosteal Flap for the Closure of Oro-antral Fistula

INTERVENTIONS:
Procedure: A Pedicled Buccal Periosteal Flap for the Closure of Oro-antral Fistula — A Pedicled Buccal Periosteal Flap for the Closure of Oro-antral Fistula

SUMMARY:
The aim of this study is to evaluate both clinically and radiologically the efficacy of using the pedicled buccal periosteal flap for closure of oroantral fistula without affecting the original intraoral anatomy.

DETAILED DESCRIPTION:
Background: Oroantral fistula (OAF) is a pathological communication between the oral cavity and the maxillary sinus. A variety of surgical techniques have been developed, with recurrence rates of up to 33%7, mainly due to wound contraction and postoperative infection. To increase the success rates of OAF closure procedures, the use of double-layered closure techniques has developed, but most of these techniques alter the original oral anatomy and may result in significant postoperative morbidity.

Purpose: The aim of this prospective study is to evaluate both clinically and radiologically the efficacy of using the pedicled buccal periosteal flap for closure of oroantral fistula without affecting the original intraoral anatomy.

Patients & Methods: Ten patients with oroantral fistula will be included in this study. The patients will be examined and managed at the Oral and Maxillofacial surgery Department, Faculty of Dentistry, Tanta University.

Preoperative evaluation: It will include the collection of demographic data, medical status and relevant history of the OAF (etiology, duration, resonance of voice, regurgitation of fluid, infection and previous surgical closure attempts). Cone beam computed tomography (CBCT) scan will be performed to determine the size of the underlying bony defect.

Surgical procedure: The buccal mucoperiosteal flap will be splitted horizontally into two layers: a deep periosteal layer and a superficial buccal mucosa layer. The fistula tract will transected at the bone level, the pedicled deep periosteal layer will be dissected and turned over the fistula at the bone level and will be stabilized using sutures. The superficial layer will be returned to its original position and sutured.

Postoperative evaluation: The patients will be evaluated clinically each week for one month regarding to healing, presence of infection, inflammation and recurrences.

ELIGIBILITY:
Inclusion Criteria:

1. patients have oroantral fistula
2. clear maxillary sinus with no infection

Exclusion Criteria:

1. Patients suffering from any systemic diseases affect healing of soft tissue
2. patients have remaining roots or foreign body in sinus indicated for cald well luc opearation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | 1 month
  0 representing no pain and 10 representing the highest level of pain
comparison of vestibular depth preoperatively and postoperatively | 1 month
  the vestibular depth measured from gingival margin to bottom of vestibule.
inflammation score scale | 1 month
  0 no inflammation, 1-3 mild inflammation,4-7 moderate inflammation,8-10 severe inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Marwa T Ibrahim, lecturer, Principal Investigator — Tanta University
Locations (1):
- Egypt, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
A Pedicled Buccal Periosteal Flap for the Closure of Oro-antral Fistula

REFERENCES:
- [Derived] Ibrahim MT, Gharieb EA, Sheta MS. A pedicled buccal periosteal flap for the closure of oro-antral fistula. BMC Oral Health. 2024 Apr 10;24(1):440. doi: 10.1186/s12903-024-04217-6. PMID 38600501